CLINICAL TRIAL: NCT04724707
Title: An Open Multicenter Observational Study (Registry) of Patients Recovered From Novel Coronavirus Infection (COVID-19) With Involvement of the Cardiovascular System or With Baseline Severe Cardiovascular Diseases
Brief Title: Russian Cardiovascular Registry of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 0509-20-2020
Record Dates: First submitted 2021-01-16; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Acute Cardiovascular Disease; Cardiovascular Diseases
Keywords: SARS-CoV-2; Covid19; Cardiovascular disease
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Samples for biochemistry, coagulation and genetic tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Myocarditis: Proven or suspected myocarditis
- Heart failure: Heart failure (NYHA functional class II-IV) before or during hospitalization with COVID-19
- ACS: Combination of COVID-19 with ACS or development of ACS during hospitalization with COVID-19 or performed percutaneous coronary intervention
- Pulmonary embolism: Proven pulmonary embolism
- Arrhythmias: Hemodynamically significant arrhythmias (atrial fibrillation, high-grade ventricular premature beats, paroxysmal ventricular arrhythmias), including those associated with the QT interval prolongation

SUMMARY:
This is a Russian multicenter observational study aimed to assess the mid-term and long-term prognosis in patients recovered from COVID-19 with the involvement of the cardiovascular system or with baseline severe cardiovascular diseases.

DETAILED DESCRIPTION:
This open multi-center observational study (registry) is designed to enroll consecutive eligible patients hospitalized with and recovered from COVID-19 (ICD-10 codes U07.1 or U07.2) with the involvement of the cardiovascular system or with baseline severe cardiovascular diseases. Data collection is ongoing for the duration of the pandemic. This study aims to assess the mid-term and long-term prognosis in this patient population. Analysis of this information may help to better predict the prognosis for patients and socio-economic burden of the coincidence of COVID-19 and cardiovascular diseases and to better inform about the optimal surveillance programs in recovered patients.

The de-identified participant data will be abstracted from the medical chart prospectively on the day of discharge or retrospectively (on the day of the first outpatient visit) and entered into an electronic database. The information will be stored in a database, and used at a later time for research studies.

Patients will be followed up for at least 12 months. Data on standard clinical assessment, echocardiography, laboratory results, assessment of the current therapy, specific cardiovascular assessment (depending on the cardiovascular disease), and outcomes will be collected, as well as additional blood samples for biomarkers substudy and central core laboratory imaging assessment (when applicable) at 3, 6 and 12 months. The investigators will contact patients by telephone to obtain information about outcomes in case of inability to visit in person.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Hospitalization with confirmed or suspected COVID-19 (ICD-10 codes U07.1 or U07.2)
3. Involvement of the cardiovascular system or baseline severe cardiovascular diseases defined as at least of the following:

   * proven or suspected myocarditis;
   * heart failure (NYHA functional class II-IV) before or during hospitalization with COVID-19;
   * combination of COVID-19 with ACS or development of ACS during hospitalization with COVID-19 or performed percutaneous coronary intervention;
   * proven pulmonary embolism;
   * hemodynamically significant arrhythmias (atrial fibrillation, high-grade ventricular premature beats, paroxysmal ventricular arrhythmias), including those associated with the QT interval prolongation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are the patients recovered from COVID-19 with the involvement of the cardiovascular system or with baseline severe cardiovascular diseases.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Death | 12 months
  Number of patients died during the follow up
Hospitalization for cardiovascular reasons | 12 months
  Number of patients hospitalized for cardiovascular reasons during the follow up
Hospitalization for any reason | 12 months
  Number of patients hospitalized for any reason during the follow up
Time to death | 12 months
  Number of days to death

SECONDARY OUTCOMES:
Mechanical support or heart transplant | 12 months
  Proportion of subjects requiring mechanical support or heart transplant during the follow up
ICD or CRT | 12 months
  Proportion of subjects requiring ICD or CRT
Quality of life | 12 months
  Changes in quality of life assessed by The Kansas City Cardiomyopathy Questionnaire (KCCQ) (scores are scaled from 0 to 100 and higher scores represent better health status and outcome)
Cardiac pacing or catheter ablation | 12 months
  Proportion of subjects requiring cardiac pacing or cathether ablation
Syncope or presyncope | 12 months
  Frequency of syncope or presyncope
Arrythmias | 12 months
  Frequency of arrythmias

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia